CLINICAL TRIAL: NCT01093430
Title: Anterior Superior Iliac Spine - A Useful Surface Anatomical Landmark for Safe and Symmetric Accessory Laparoscopic Port Entry
Brief Title: Is the Anterior Superior Iliac Spine a Useful Landmark at Laparoscopy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Free Hampstead NHS Trust (Other)
Responsible Party: Dr. Adam Magos,. Consultant Gynaecologist/Honorary Senior Lecturer, Royal Free Hospital, Hampstead, London NW3 2QG, UK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AM2009/1
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Surgical Techniques; Laparoscopy
Keywords: Gynecological surgery; laparoscopic ports; neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior superior iliac spine (Experimental): The position of the right and left laparoscopic port sites will be determined by palpation of the nearby anterior superior iliac spine of the pelvic bone.
  Interventions: Procedure: Anterior superior iliac spine
- Control (Active Comparator): The position of the right and left laparoscopic port sites will be determined by visual inspection of the anterior abdominal wall.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Anterior superior iliac spine — The position of the right and left laparoscopic port sites will be determined by palpation of the nearby anterior superior iliac spine of the pelvic bone.
  Other Names: Bony landmark
  Arms: Anterior superior iliac spine
Procedure: Control — The position of the right and left laparoscopic port sites will be determined by visual inspection of the anterior abdominal wall.
  Other Names: Visual
  Arms: Control

SUMMARY:
The purpose of this study is to study port symmetry and the incidence of anterior abdominal wall neuropathy associated with gynaecological surgery.

DETAILED DESCRIPTION:
We plan to study patients undergoing gynaecological laparoscopy. Patients will be randomized to two techniques for determining where to position the right and left lateral laparoscopic ports, and port symmetry will be assessed at the end of surgery. We also plan to study patients undergoing any type of gynaecological surgery to determine the incidence of sensory neuropathy involving the lower abdomen according to the route of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Due to undergo elective gynaecological surgery, including laparoscopy

Exclusion Criteria:

* Previous laparoscopy
* Junior intern as primary surgeon

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Symmetry of lateral laparoscopic ports | On the completion of laparoscopy and before the general anaesthetic is reversed
  The precise location in the horizontal and vertical planes of the right and left lateral port sites will be measured to assess port symmetry.

SECONDARY OUTCOMES:
Neuropathy | Before, immediately after and 2 weeks after gynaecological surgery
  Evidence of ilio-hypogastric and ilio-inguinal neuropathy will be sought at the above time frames.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Magos, MD FRCOG, Principal Investigator — Royal Free Hamsptead NHS Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom